CLINICAL TRIAL: NCT05487170
Title: A Phase 1/2, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Chaperone-mediated Protein Degrader RNK05047 in Subjects With Advanced Solid Tumors (CHAMP-1)
Brief Title: A Study of RNK05047 in Subjects With Advanced Solid Tumors/Diffuse Large B-cell Lymphoma (CHAMP-1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ranok Therapeutics (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ranok Therapuetics Co. Ltd. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RNK05047-01
Record Dates: First submitted 2022-07-12; First posted 2022-08-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; DLBCL
Keywords: protein degrader

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RNK05047 (Experimental): Dose-escalation of RNK05047 IV infusion
  Interventions: Drug: RNK05047

INTERVENTIONS:
Drug: RNK05047 — RNK05047 is a chaperone-mediated protein degrader administered as IV infusion once weekly for 3 consecutive weeks in a 4-week cycle (no treatment in the fourth week).

SUMMARY:
This is a first in human, Phase 1/2 open-label multi-center, dose escalation and expansion study to evaluate the safety, tolerability, PK, PD and efficacy of RNK05047 when administered an intravenous (IV) infusion to subjects with advanced solid tumors, including diffuse large B-cell lymphoma (DLBCL).

This is a 2-part study (dose escalation, cohort expansion) with sequential enrollment.

DETAILED DESCRIPTION:
In Part 1, enrolled subjects will receive IV RNK05047 once weekly for 3 consecutive weeks in a 4-week cycle (no treatment in the fourth week). The dose-escalation phase will follow a standard 3+3 design, with 3 subjects enrolled into the first dosing cohort to receive RNK05047 at the starting dose of 0.75 mg/kg.

In Part 2, once RP2D has been established, additional subjects (3 to 5 cohorts of approximately 15 subjects per cohort) will be enrolled in the cohort-expansion phase of the study. Tumor types for these cohorts will be determined based on data from the dose-escalation phase of the study and emerging results from preclinical studies or other scientific data. These dose expansion cohorts in all groups may be done concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented locally advanced or metastatic solid tumor
* Refractory or intolerant to all available standard-of-care therapies for advanced disease
* Measurable disease
* Archived tumor tissue collected
* ECOG Performance Status of 0 or 1
* BMI ≥ 18 kg/m2
* Adequate liver, renal, hematologic, and coagulation parameters
* Negative serum pregnancy test (for women of childbearing potential) at Screening and a negative urine or serum pregnancy test on Day 1 prior to the first infusion
* Males and females of childbearing potential must agree to use a highly effective method of contraception during treatment and for at least 4 months after the last dose of study treatment.
* Must be able to understand and comply with the conditions of the protocol and must have read and understood the consent form and provided written informed consent.

Exclusion Criteria:

* Concurrent anticancer therapy: Radiotherapy, chemotherapy, biological therapy, or other anticancer investigational agents NOTE: at least 5 half-lives must have been ensued for any prior systemic cancer therapy agent before subject received the study drug on Day 1
* Unresolved toxicities from prior anticancer therapy, defined as not having resolved according to CTCAE version 5.0 Grade ≤ 1, excluding Grade 1 alopecia
* Presence or suspicion of active central nervous system (CNS) metastases and/or leptomeningeal carcinomatosis
* Peripheral neurotoxicity ≥ Grade 2 according to CTCAE v5.0
* Known active infection with HIV, HTLV-1, hepatitis B or C
* Women who are pregnant or breastfeeding
* History of another malignancy unless the subject has been treated with curative intent for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of DLTs | through 1 cycle/4 weeks
Part 1: Incidence of TEAEs | through study completion, an average of 1 year
Part 2: Incidence of TEAEs | through study completion, an average of 1 year
Part 2: Objective response rate (ORR) based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 2: Duration of response (DoR) based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 2: Progression-free Survival (PFS) based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 2: Disease Control Rate (DCR) based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Part 1: Plasma concentration RNK05047 | Through Cycle 3/approximately 12 weeks
Part 1: ORR based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 1: DoR based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 1: PFS based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 1: DCR based on RECIST 1.1/RECIL 2017 | through study completion, an average of 1 year
Part 2: Plasma concentration RNK05047 | Through Cycle 3/approximately 12 weeks
Part 2: Overall Survival (OS) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Linda Grummer, Study Director — Ranok Therapeutics
Locations (5):
- United States (3):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Weill Cornell - NY Presbyterian Hospital, New York, New York
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No